CLINICAL TRIAL: NCT04078542
Title: Assessing Prevalence and Main Features of Chronic Refractory Cough in Different Specialist Settings.
Brief Title: Prevalence and Main Features of Chronic Refractory Cough.
Acronym: ASSESS-CRC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Raffaele Antonelli Incalzi, Full Professor of Internal Medicine, Campus Bio-Medico University
Other Study IDs: ComEtx
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic cough: Subject complaining cough from at least 8 weeks

SUMMARY:
Cough is among the most common causes of medical consultation in primary care.[1] Chronic cough, arbitrarily defined as symptom persisting more than 8 weeks, has been variably reported in different settings and geographical area, with an overall prevalence of 10-20% in the general population, that increases up to 40-50% in pneumology specialist clinics.[2,3] While acute cough is generally caused by the common cold and typically lasts one to three weeks, chronic persisting cough can underlie more serious disease processes. Moreover, it can impair quality of life,[4] possibly leading to tiredness, urinary incontinence, and eventually syncope. It also has psychosocial effects such as embarrassment and negative impact on social interactions.

A careful clinical history may provide important diagnostic clues that allow therapeutic trials without the need of further investigations.[5] Smoking history, medication list and presence and character of sputum should be carefully detailed. Identification of the causes of productive cough is generally straightforward and strategies for intervention and treatment are well defined.[5] Conversely, chronic dry or poorly productive cough represents a greater diagnostic challenge. Several studies have shown that in nonsmokers with normal chest radiography who are not taking ACE-inhibitor, chronic cough is usually due to asthma, rhinosinusitis or gastro-esophageal reflux (GER).[6] Many dedicated algorithms have been identified to guide the diagnostic phase and to sequentially coordinate the execution of further diagnostic deepening and/or empirical treatments, based on cost-effectiveness principles.[5,7-9] Among these, the European Respiratory Society (ERS) recommendations[5] are widely applied in clinical practice and broadly parallel those released by the American College of Chest Physicians[7]. This notwithstanding, a proportion of cases do not reach a definite diagnosis and resolutive treatment[7]. This condition is termed chronic refractory cough (CRC), chronic idiopathic cough, or unexplained chronic cough.[7,10] It can be diagnosed when patients have no identified causes of chronic cough (unexplained or idiopathic chronic cough) or when the cough persists after investigation and treatment of cough-related conditions. Because patients with unexplained chronic cough often receive specific therapies, such as inhaled corticosteroids or proton pump inhibitors, they can also be classified as having CRC.

The real prevalence of CRC is not well-know and many cases of CRC may be actually misdiagnoses due an incomplete application of recommended work-up. In the present study we aim to estimate the prevalence of chronic cough in different care settings, together with the prevalence of CRC according to a systematic and integrated approach. The careful application of the recommendation defined by ERS guidelines will allow to detect truly refractory cases of chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* complaining chronic cough (lasting more than 8 weeks)

Exclusion Criteria:

* Unwilling to participate

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be screened for the presence of cough and those complaining chronic cough (i.e. lasting more than 8 weeks) will be included. Only subjects aged less than 18 years will be excluded and no other specific exclusion criteria will be adopted, in order to gather data on a real life population.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients complaining cough lasting more than 8 weeks during geriatric and respiratory specialist visits | 2 years
  to estimate the prevalence of chronic cough in different settings, i.e. in geriatric and in pneumology specialist clinics
Proportion of patients with chronic refractory cough on all patients with chronic cough coming to medical attention during geriatric or respiratory specialist visits | 2 years
  to estimate the prevalence of chronic refractory cough (CRC) in subject with chronic cough - CRC will be diagnosed if cough persists despite guideline based management - In particular, CRC will be defined as cough persisting after a complete diagnostic work-up and despite extended trials of empirical therapy.
describe the clinical and demographic characteristics (age, sex, comorbidities, smoke hystory, type of cough presentation, educational level) of patients with chronic refractory cough | 2 years
  to define patient's socio-demographical and clinical characteristics associated with the diagnosis of chronic refractory cough

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, MD, Principal Investigator — Campus Bio Medico
Locations (3):
- Italy (3):
  - Campus Bio-Medico di Roma, Roma
  - IRCCS Maugeri Tradate, Roma
  - Policlinico Universitario Agostino Gemelli Università Cattolica del Sacro Cuore, Roma

IPD SHARING:
Plan to Share IPD: No